CLINICAL TRIAL: NCT03205410
Title: Remote Ischemic Preconditioning as a New Method of Nephroprotection in Patients Undergoing Cardiac Surgery
Brief Title: Remote Ischemic Preconditioning as a New Method of Nephroprotection
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medical University of Lodz (Other)
Responsible Party: Principal Investigator, Karolina Stokfisz, M.D., Medical University of Lodz
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: RNN/286/13/KE
Record Dates: First submitted 2017-06-29; First posted 2017-07-02 (Actual); Last update posted 2017-07-02 (Actual); Status verified 2017-06

CONDITIONS: Acute Kidney Injury
Keywords: remote ischemic preconditioning; cardiac surgery-associated acute kidney injury; neutrophil gelatinase-associated lipocalin
MeSH Terms: conditions — Acute Kidney Injury

STUDY DESIGN:
Who Masked: Investigator
Masking Description: Patients were randomly assigned in 1:1 ratio to either the RIPC group or the control group by means of a computerized randomization table.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Patients with RIPC (Experimental): intervention: remote ischemic preconditioning - three cycles of 5-min ischemia, achieved by inflation of blood-pressure cuff to 200 mmHg, followed by 5-min reperfusion while the cuff was deflated were applied to the upper left arm.
  Interventions: Procedure: remote ischemic preconditioning
- Patients without RIPC (Sham Comparator): intervention: no - remote ischemic preconditioning - in controls, the cuff was placed around the arm but not inflated.
  Interventions: Procedure: no - remote ischemic preconditioning

INTERVENTIONS:
Procedure: remote ischemic preconditioning — The remote ischemic preconditioning protocol described before began after anesthesia induction, and was completed prior to the start of surgery.
  Other Names: RIPC
  Arms: Patients with RIPC
Procedure: no - remote ischemic preconditioning — The sham - remote ischemic preconditioning protocol described before began after anesthesia induction, and was completed prior to the start of surgery.
  Other Names: no-RIPC
  Arms: Patients without RIPC

SUMMARY:
Remote ischemic preconditioning (RIPC), elicited by brief episodes of ischemia and reperfusion in distant tissue, offers a protection against acute kidney injury (AKI) in patients after cardiac surgery. Investigators conducted a prospective, randomized, controlled clinical trial to assess whether RIPC reduces the incidence of AKI measured by standard way using serum creatinine concentration (SCr) and with use of serum level of neutrophil gelatinase-associated lipocalin (NGAL) as a new potential biomarker of a kidney injury. Moreover the aim of investigation was to analyse the safety and clinical outcomes of RIPC after elective, isolated, primary off-pump coronary artery bypass graft surgery (OPCAB).

DETAILED DESCRIPTION:
Cardiac surgery patients have a high risk of AKI. The development of AKI is associated with higher mortality and a higher risk for complications in patients undergoing cardiac surgery. However, there are no effective clinical strategies for preventing prevalence of AKI. RIPC as a simple, inexpensive way of protecting tissues against ischemic damage, may also reduce kidney injury. That makes RIPC under the area of interests of many researches which apply this method to prevent AKI. Investigators conducted a single-center, double-blind trial involving patients at high risk of postoperative AKI, in which want to check wether RIPC reduce the prevalence of AKI, according Kidney Disease: Improving Global Outcomes (KDIGO) definition, by increase in SCr. Furthermore researchers want to investigate a benefit from RIPC in reduction of level of SCr and higher glomerular filtration rate (GFR) 72 hours after off-pump coronary artery bypass as well as reduction of postoperative expression of NGAL an early biomarker of AKI.

ELIGIBILITY:
Inclusion Criteria:

* Human patients with coronary artery disease.

Exclusion Criteria:

* history of cardiac surgery,
* acute myocardial infarction up to 7 days before surgery,
* chronic kidney disease in 4th or 5th stadium (eGFR<30 ml/min/1,73m2),
* peripheral vascular disease affecting upper limbs,
* history of severe injuries and surgeries in 2 months before cardiac surgery,
* history of cancer, acute inflammation during hospitalization,
* chronic autoimmunology diseases,
* dialysis patients.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2014-01-01 (Actual); Primary Completion 2014-12-31 (Actual); Study Completion 2014-12-31 (Actual)

PRIMARY OUTCOMES:
incidence of acute kidney injury within 72 hours after cardiac surgery | 72 hours after cardiac surgery
  increase in serum creatinine level by more than 50% or more than 0.3mg/dL from baseline within 72 h after surgery
NGAL level | 3 hours after cardiac surgery
  increased NGAL level within 3 hours after cardiac surgery

SECONDARY OUTCOMES:
length of hospitalization | through hospitalization completion, an average of 14 days
  time until discharge from the hospital
length of intensive care unit (ICU) stay | through ICU stay completion, an average of 5 days
  time until discharge from ICU
ventilation time | through ICU stay completion, an average of 5 days
  time of mechanical ventilation
occurrence of postoperative atrial fibrillation | through ICU stay completion, an average of 5 days
  incidence of atrial fibrylation in continous electrocardiogram registration
time of renal replacement therapy | through ICU stay completion, an average of 5 days
  days of renal replacement therapy
death | from date of randomization until the date of death from any cause, assessed up to 2 years
  death from any cause

CONTACTS AND LOCATIONS:
Overall Officials: Marzenna Zielinska, MD,PhD,Prof., Study Chair — Medical University of Lodz
Locations (1):
- Intensive Cardiac Therapy Clinic, Lodz, Poland

IPD SHARING:
Plan to Share IPD: Yes
The datasets used and/or analyzed during the current status of the study are available from the corresponding author on reasonable request.

REFERENCES:
- [Derived] Stokfisz K, Ledakowicz-Polak A, Zagorski M, Jander S, Przybylak K, Zielinska M. The clinical utility of remote ischemic preconditioning in protecting against cardiac surgery-associated acute kidney injury: A pilot randomized clinical trial. Adv Clin Exp Med. 2020 Feb;29(2):189-196. doi: 10.17219/acem/112610. PMID 32091672